CLINICAL TRIAL: NCT03390348
Title: An In-home Observational Study to Compare Infant Crying and Fussing Parameters Documented by the LENA Recorder With Those Documented Via Parental E-diaries
Acronym: LENUS
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: LENA Foundation (Unknown); ObvioHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: OBVIO-DAN-001; EBB17GC16811 (Other: DAPH)
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Crying; Fussy Infant (Baby)
MeSH Terms: conditions — Crying

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LENA Recorder — Use of the LENA recorder to document crying and fussing

SUMMARY:
This is a in-home observational study of 12 healthy term infants of ≤15 weeks of age to compare infant crying and fussing parameters documented by the LENA recorder with those documented via parental e-diaries

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants, age ≤15 weeks
* Singleton infants (≥37 and ≤42 weeks gestation)
* Birth weight within normal range for gender and gestational age
* Informed consent from parent or legal guardian whose age is ≥18 years old
* Live in a household with reliable electronic communication capability (e.g. smart phone, computer, internet access)
* Infants who are breastfed and/or are consuming any commercial infant formula as a major nutrient source
* Parent's/guardian's English literacy sufficient to follow instructions and complete forms

Exclusion Criteria:

Infants:

* Currently or within last 30 days prior to screening, participation in any other investigational studies
* Known to have current or previous illness/condition which could interfere with the study outcome, as per Investigator's clinical judgment

Parents/Guardians of infants:

* Known to have a significant medical condition (including during pregnancy) that might interfere with the study, as per Investigator's clinical judgment
* Inability to comply with study protocol, as per the Investigator's judgement

Max Age: 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term infants of ≤15 weeks of age
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Comparison of the crying and fussing documented by the LENA recorder with the crying and fussing documented in the parental e-diaries | 14 days
  Comparison of the crying and fussing documented by the LENA recorder with the crying and fussing documented in the parental e-diaries

SECONDARY OUTCOMES:
Quantification of inconsolable and unexplainable crying and fussing times based on parental e-diaries | 14 days
  Quantification of inconsolable and unexplainable crying and fussing times based on parental e-diaries
Quantification of inconsolable and unexplainable crying and fussing times detected by the LENA recorder | 14 days
  Quantification of inconsolable and unexplainable crying and fussing times detected by the LENA recorder

OTHER OUTCOMES:
Using a parental questionnaire, investigate the usability of the e-diary and ClaimIt app interface | 14 days
  Using a parental questionnaire, investigate the usability of the e-diary and ClaimIt app interface
Using a parental questionnaire, investigate the usability of the LENA recording device | 14 days
  Using a parental questionnaire, investigate the usability of the LENA recording device
Explore possible correlations between crying and fussing behaviors and infant diet reports | 14 days
  Explore possible correlations between crying and fussing behaviors and infant diet reports

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — Obvio Health
Locations (1):
- ObvioHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dykstra JR, Sabatos-Devito MG, Irvin DW, Boyd BA, Hume KA, Odom SL. Using the Language Environment Analysis (LENA) system in preschool classrooms with children with autism spectrum disorders. Autism. 2013 Sep;17(5):582-94. doi: 10.1177/1362361312446206. Epub 2012 Jul 2. PMID 22751753
- [Result] Canault M, Le Normand MT, Foudil S, Loundon N, Thai-Van H. Reliability of the Language ENvironment Analysis system (LENA) in European French. Behav Res Methods. 2016 Sep;48(3):1109-24. doi: 10.3758/s13428-015-0634-8. PMID 26174716